CLINICAL TRIAL: NCT07254949
Title: Vision and Proprioception Evaluation With Robotics After Stroke
Acronym: VIPERS
Status: Not yet recruiting | Type: Observational
Sponsor: Dr. Sean Dukelow (Other)
Responsible Party: Sponsor-Investigator, Dr. Sean Dukelow, Principal Investigator, University of Calgary
Organization: University of Calgary (Other)
Other Study IDs: REB25-1170; 197953 (Other Grant/Funding Number: Canadian Institutes of Health Research)
Record Dates: First submitted 2025-11-19; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Stroke; Control Condition
Keywords: Stroke; Sensation; Movement; Vision; Robotics; Eye-Tracking; Imaging
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Stroke: Stroke Participants - Individuals with first time stroke
- Control: Control Participants - Individuals not suffering stroke or other neurological disorders

SUMMARY:
Stroke is highly prevalent in Canada and can lead to profound upper limb impairments in motor and sensory function, as well and vision. Clinical assessments for these functions often lack sensitivity making detecting impairments and tracking their recovery after stroke difficult. It is known that sensory function and vision interact to inform motor behaviours, yet how each of these modalities might contribute to motor impairments and subsequent recovery after stroke is undetermined.

Using robotics to assess neurologic function after a stroke can be very beneficial, as they can measure on the scale of millimetres and milliseconds which can more easily detect subtle deficits in a persons function. Compared to current clinical tools, robotics offer greater objectivity and reliability, as they do not rely on the examiners clinical experience and/or impression. The use of robotics not only offers a more precise measurement, but robotics assessments can be completed in a relatively short amount of time, in comparison to some of the current clinical assessment tools, which can take along time to complete. In addition to robotics, collecting neuroimaging (MRI/CT) will allow us to relate our robotic and eye-tracking measures to neuroanatomical information about the person's stroke. With this data, we will assess how the brain changes post-stroke in relation to the recovery of motor, sensory and visual functions.

This research will: 1) examine the relationship between visual and proprioceptive impairment on motor and eye movement behaviour over time after stroke, and 2) identify neuroanatomical correlates of visual, proprioceptive and sensory integrative dysfunction that impact motor recovery after stroke and examine the ability of regional damage and network disruption to predict recovery.

Objectives:

1. Determine the impact of visual field loss and visual neglect in stroke survivors with impaired movement over the first 6 months post-stroke.
2. Identify the impact of Proprioceptive Impairment and Sensory Integration Impairment on recovery post-stroke using robotics and eye tracking.
3. Understand the impact of damage to neuroanatomic structures involved in vision, proprioception and sensory integration on motor recovery using MRI after stroke.

The VIPERS study is recruiting both stroke and control participants. Stroke participants are recruited within the first 28 days post-stroke and are assessed longitudinally across the first 6-months post-stroke (four study timepoints). Control participants just complete a single session.

ELIGIBILITY:
Inclusion criteria for stroke participants:

* 18 years of age or older
* First clinical diagnosis of stroke
* No recent muscle skeletal injuries to the arms, neck, or back
* No history of other neurological disease/injury (Ie. MS, Parkinson's, Brain Tumour, etc.)
* Corrected vision 20/50 or better
* Able to follow multi-step commands.
* Living independently prior to stroke
* Can consent to participate in research

Inclusion criteria for control participants:

* 18 years of age or older
* No history stroke, or Trans Ischemic Attack (TIA)
* No recent muscle skeletal injures to the arms, neck, or back
* No history of other neurological disease/ injury (Ie. MS, Parkinson's, Brain Tumour, etc)
* No pre-stroke history of eye movement disorders
* Corrected vision 20/50 or better
* Able to follow multi-step commands
* Can consent to participate in research

Exclusion Criteria:

* Prior history of stroke/significant neurologic problem (e.g. Parkinson's)
* Symptomatic medical conditions that would interfere with participation (e.g. uncontrolled angina)
* Contraindications to Magnetic Resonance Imaging (MRI)
* Pre-stroke history of visual field/oculomotor abnormalities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 425 participants will be recruited for this study (225 stroke participants and 200 matched control participants who have not experienced a stroke). All participant will be aged 18 or older.
Sampling Method: Non-Probability Sample
Enrollment: 425 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2031-01 (Estimated); Study Completion 2031-06 (Estimated)

PRIMARY OUTCOMES:
Visually Guided Reaching Score | Enrolment to six-months post stroke

OTHER OUTCOMES:
Visually Guided Reaching Score (no vision) | Enrolment to six-months post stroke
Proprioceptive Saccade task scores | Enrolment to six-months post stroke
Arm Movement Matching (vision) | Enrolment to six-months post stroke
Arm Movement Matching | Enrolment to six-months post stroke
Arm position matching (vision) | Enrolment to six-months post stroke
Arm Position Matching Score | Enrolment to six-months post stroke
Visually Guided Reaching Score | From enrolment to six-months post stroke
Anti-saccade task score | Enrolment to six-months post stroke
Pro-saccade task score | Enrolment to six-months post-stroke
Behavioural Inattention Test (BIT) | Enrolment to six-months post-stroke
Visual Impairment Screening Assessment (VISA) | Enrolment to six-months post-stroke
Humphrey's Visual Field Analyzer (VFA) | Enrolment to six-months post stroke
Thumb Localization Test (TLT) | Enrolment to six-months post stroke
Medical Research Council Strength Scale | Enrolment to six-months post stroke
Modified Ashworth Scale (MAS) | Enrolment to six-months post stroke
Fugl-Meyer Assessment-Upper Extremity (FMA-UE) | Enrolment to six-months post stroke
Functional Independence Measure (FIM) | Enrolment to six-months post stroke

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Carewest Dr. Vernon Fanning Centre, Calgary, Alberta
  - Foothills Medical Centre, Calgary, Alberta

IPD SHARING:
Plan to Share IPD: No
Formal data transfer agreements/legal contracts are required to share IPD with other researchers outside of the main study site.